CLINICAL TRIAL: NCT00591708
Title: Calcium Metabolism in Asian Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Berdine Martin, Research Scientist, Nutrition Science, Purdue University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: AR40553; R01AR040553 (NIH)
Record Dates: First submitted 2007-12-26; First posted 2008-01-11 (Estimated); Last update posted 2018-05-09 (Actual); Status verified 2018-05

CONDITIONS: Bone Mineralization; Adolescent Development
Keywords: calcium; bone; bone density; adolescence
MeSH Terms: interventions — calcium citrate malate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- B (Experimental): Supplementation of a higher level of calcium (500-1300 mg/d) via calcium fortified beverages (calcium citrate malate) to a basal diet of 600 mg/d for 21 consecutive days. All excreta will be collected.
  Interventions: Dietary Supplement: Beverage fortified with calcium citrate malate
- A (Experimental): Supplementation of a lower level of calcium (0-400 mg/d) via calcium fortified beverages (calcium citrate malate) to a basal diet of 600 mg/d for 21 consecutive days. All excreta will be collected.
  Interventions: Dietary Supplement: Beverage containing calcium citrate malate

INTERVENTIONS:
Dietary Supplement: Beverage containing calcium citrate malate — Beverages containing a lower amount of calcium (0-400 mg/d) will be supplemented to a basal diet containing 600 mg/d Ca. The controlled diet will be consumed for 21 consecutive days.
  Arms: A
Dietary Supplement: Beverage fortified with calcium citrate malate — Beverages containing a higher amount of calcium (500-1300 mg/d) will be supplemented to a basal diet containing 600 mg/d Ca. The controlled diet will be consumed for 21 consecutive days.
  Arms: B

SUMMARY:
Maximizing calcium retention by the skeleton within the genetic potential is a key strategy to prevent osteoporosis. It has been shown that calcium retention varies between blacks and whites and between gender within race. This study is designed to study the relationship between calcium intakes and calcium retention in Asian adolescent girls and boys. It is hypothesized that calcium intakes which maximize calcium retention will be lower in Asians than for whites studies under the same conditions. In addition it is thought that the differences between races in the physiological mechanisms involved in calcium metabolism will result in a lower calcium intake required to observe a plateau in calcium retention. This is turn could be translated into lower calcium requirements in Asians relative to Caucasians for achieving optimal peak bone mass.

DETAILED DESCRIPTION:
Adolescent Asian boys and girls will consume a controlled diet for two three-week periods. The basal diet will contain 600 mg/d calcium and will be supplemented with beverages fortified with calcium citrate malate to achieve a range of intakes from 600-2100 mg Ca/d. Each participant will be studied on one of four combinations of a lower and a higher calcium intake within that range in a cross-over design.

ELIGIBILITY:
Inclusion Criteria:

* healthy teens of Asian descent

Exclusion Criteria:

* malabsorptive disorders
* anemia
* smoking, illegal drugs
* oral contraceptives
* pregnancy
* drugs that influence calcium metabolism
* body weight for height greater than 85 percentile

Ages: 11 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2004-07; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Calcium retention (mg/d) | Metabolic balance will be determined over a two week period on a controlled diet after equilibration for one week on the same diet.

SECONDARY OUTCOMES:
Serial serum biochemistry profiles (PTH, 1,25 dihydroxy-vitamin D, calcium) | Six serial measurements in 10 hours after ingestion of a calcium load representing one third of the daily consumption

CONTACTS AND LOCATIONS:
Overall Officials: Connie Weaver, PhD, Principal Investigator — Department of Foods and Nutrition, Purdue University; Berdine R Martin, PhD, Study Director — Department of Foods and Nutrition, Purdue University
Locations (1):
- Department of Foods and Nutrition, Purdue University, West Lafayette, Indiana, United States

REFERENCES:
- [Derived] Wu L, Martin BR, Braun MM, Wastney ME, McCabe GP, McCabe LD, DiMeglio LA, Peacock M, Weaver CM. Calcium requirements and metabolism in Chinese-American boys and girls. J Bone Miner Res. 2010 Aug;25(8):1842-9. doi: 10.1002/jbmr.76. PMID 20205166